CLINICAL TRIAL: NCT02901600
Title: Modification of the Expression and the Localization of DMBT1 (Deleted in Malignant Brain Tumor 1) in Colorectal Cancer
Brief Title: Expression of DMBT1 in Colorectal Cancer Patients
Acronym: DMBT1
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RT-06
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: DMBT1 Protein, Human; Colorectal Cancer
Keywords: DMBT1 expression; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with colorectal cancer: Fresh tissue samples from individuals with colorectal carcinoma taken from the tumor as well as from resection margins will be used for the detection of a potential marker of carcinogenesis.
  Interventions: Other: Detection of the expression of DMTB1 by immunohistochemistry
- Patients with adenomatous polyps: Fresh tissue samples from individuals with adenomatous polyps will be used for the detection of a potential marker of carcinogenesis.
  Interventions: Other: Detection of the expression of DMTB1 by immunohistochemistry
- Control patients: Fresh tissue samples from individuals without colorectal carcinoma will be used as control.
  Interventions: Other: Detection of the expression of DMTB1 by immunohistochemistry

INTERVENTIONS:
Other: Detection of the expression of DMTB1 by immunohistochemistry

SUMMARY:
Although colorectal cancer is a preventable and curable disease if early stage tumors are removed, it is still the fourth cause of cancer worldwide and the second leading cause of death in many industrialized countries. The 5-year survival is about 55% often due to a late detection. Then, the identification of sensitive and specific molecular markers is therefore a major challenge for early diagnosis and prognosis of this disease.

Preliminary work have reported variations in the expression of DMBT1 (deleted in malignant brain tumor 1), a glycoprotein co-secreted with mucins in the light of the glands, during several stages of colon carcinogenesis. The goal of this study is to study by mass spectrometry (MS), alterations in the repertoire of glycosylation of mucins from colorectal tumors of various stages, grades, and recurrence status.

ELIGIBILITY:
Inclusion Criteria:

* for colon cancer: patients surgically treated for colorectal cancer at the Group of hospitals of the Catholic Institute of Lille.
* for adenomatous polyps : patients treated for adenomatous polyps at the Group of hospitals of the Catholic Institute of Lille.
* for controls: patients surgically treated for diverticular disease at the Group of hospitals of the Catholic Institute of Lille.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with colorectal carcinoma, with polyps or without colonic pathology
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Semi-quantitative determination of the histological expression of DMBT1 | at baseline
  The expression of DMTB1 will be determined by observation of the slides after immunohistochemistry using an anti-DMBT1 antibody
Determination of the histological localisation of DMBT1 | at baseline
  The localisation of DMTB1 will be determined by observation of slides after immunohistochemistry using an anti-DMBT1 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Mihalache, MD, PhD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No